CLINICAL TRIAL: NCT01260987
Title: Conventional Versus Fractional CO2 Laser Assisted Photodynamic Therapy for Basal Call Carcinomas and Actinic Keratoses
Brief Title: Fractional CO2 Laser Assisted Photodynamic Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Christina Haak, MD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-1-2010-044; 2010-020179-22 (EudraCT Number)
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Actinic Keratosis; Basal Cell Carcinoma
Keywords: Moderate to severe actinic keratoses; Difficult to treat nodular basal cell carcinomas
MeSH Terms: conditions — Keratosis, Actinic; Carcinoma, Basal Cell

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AK split-face treatment (Active Comparator): Split-face treatment of two symmetrical areas with moderate to severe actinic keratoses. One area is treated with conventional PDT the other with fractional laser assisted PDT.
  Interventions: Drug: Conventional photodynamic therapy; Drug: Fractional CO2 laser assisted PDT
- Fractional laser assisted PDT for BCC (Active Comparator): Difficult to treat nodular basal cell carcinomas in the face is pretreated with fractional CO2 laser followed by methyl-aminolevulinate PDT.
  Interventions: Drug: Fractional CO2 laser assisted PDT
- Konventional PDT for BCC (Active Comparator): Difficult to treat nodular basal cell carcinomas in the face is treated with methyl-aminolevulinate PDT.
  Interventions: Drug: Conventional photodynamic therapy

INTERVENTIONS:
Drug: Conventional photodynamic therapy — Photodynamic therapy using methyl-aminolevulinate and red light (37 J/cm2)
  Arms: AK split-face treatment; Konventional PDT for BCC
Drug: Fractional CO2 laser assisted PDT — Pretreatment with fractional CO2 laser before methyl-aminolevulinate PDT
  Arms: AK split-face treatment; Fractional laser assisted PDT for BCC

SUMMARY:
Nodular Basal Cell Carcinomas:

Compare the efficacy and safety of conventional versus fractional laser assisted PDT for difficult to treat nodular cell carcinomas in the face.

Actinic keratosis:

Compare the efficacy and safety of conventional versus fractional laser assisted PDT for moderate to severe actinic keratoses located in the face and on the hands.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Skin type I-III
* Fertile women using secure birth control
* Moderate to severe actinic keratoses in the face or on the hands,
* Difficult to treat nodular basal cell carcinomas in the face

Exclusion Criteria:

* Pregnancy or breast feeding patients
* Patients with porphyria
* Patients with Gorlins syndrome
* Patients with a tendency to produce hypertrophic scars or keloids
* Patients with known allergy to Metvix
* Patients who are not considered able to follow the treatment protocol (e.g. severely alcoholic, dementia, mentally ill etc.)
* Patients with pigmented or morphea basal cell carcinomas
* Know herpes simplex virus infection in treatment areas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Treatment response | 3 months
  Clinical evaluation by a blinded physician.
Reoccurrence | 12 months
  Clinical evaluation by a blinded physician
Treatment response | 12 months
  Blinded histological examination from patients with basal cell carcinomas

SECONDARY OUTCOMES:
Pain | during laser and PDT
  Patient score (VAS 0-10)
Adverse effects | 12 months
  scaring, hyper- and hypopigmentation
Fluorescence | 3 hours
  Methyl-amonolevulinate uptake
Cosmetic result | 12 months
  4-point scale

CONTACTS AND LOCATIONS:
Overall Officials: Merete Hædersdal, PhD,DrMedSci, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Department of Dermatology, Bispebjerg Hospital, Copenhagen, Denmark